CLINICAL TRIAL: NCT05570955
Title: Deucravacitinib Adherence Study
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: IRB00087852
Record Dates: First submitted 2022-09-22; First posted 2022-10-07 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Psoriasis
MeSH Terms: conditions — Psoriasis

STUDY DESIGN:
Intervention Model Description: All participants will receive their medication with electronic monitors attached. 50% of those enrolled will receive reminders to take their medication the other 50% will not.
Who Masked: Participant
Masking Description: Participants will not be told that the monitors attached to their medication is recording their usage
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Other): 50% of subjects will be randomized to a reporting tool designed to promote better adherence to treatment by having subjects report their progress on a weekly basis (the goal is not to test this tool but to help assure there is a broad range of adherence behavior including some positive adherence outliers)
  Interventions: Behavioral: Text reminder
- No Intervention (No Intervention): 50% of subjects will not receive additional outreach to improve adherence

INTERVENTIONS:
Behavioral: Text reminder — weekly text to remind use of drug
  Arms: Intervention

SUMMARY:
Psoriasis patients are very poorly adherent to topical treatment. If adherence issues are ignored, poor adherence may limit the real-world efficacy of deucravacitinib, too. Forty psoriasis patients recruited from Wake Forest Baptist Health Dermatology Clinic will be enrolled. Twenty will be randomized to a reporting intervention designed to promote better adherence and the remaining 20 patients will serve as controls who will not receive a reporting intervention. Through qualitative interviews of the 40 patients recruited, we plan to study the behaviors of the most adherent patients to better understand specific beliefs and behaviors of adherent patients and to identify practical, modifiable factors that can improve adherence. We will also compare treatment outcomes and efficacy of deucravacitinib between the most and least adherence patients.

DETAILED DESCRIPTION:
STUDY OBJECTIVES

* PRIMARY OBJECTIVE: The primary objective of the proposed study is to identify adherence outliers (high and low adherence), specific beliefs, and behaviors that correspond to better and worse adherence to oral treatment of psoriasis.
* SECONDARY OBJECTIVE: The investigators will study the efficacy and safety of deucravacitinib in patients who are highly adherent to treatment compared to patients who do not take the medication as directed (including both those who undertreat and overtreat).

  * Safety endpoints will include reported adverse events.
  * For the characterization of adherence to deucravacitinib, adherence endpoints will include the proportion of subjects with 80% or greater adherence, days with missed treatment, days with overuse, and premature discontinuation.

ELIGIBILITY:
Inclusion Criteria:

* Patients with moderate-to-severe plaque psoriasis. Standard criteria for moderate-to-severe plaque psoriasis will be used (BSA greater than or equal to 3% or face/palm/sole/genital involvement or severe effect on Quality of Life).
* Subject must be 18 years of age or older.
* Subject must have a working knowledge of English.
* Approved birth control methods required for females of childbearing potential.
* Baseline TB test.

Exclusion Criteria:

* Patients without a diagnosis of moderate-to-severe plaque psoriasis.
* Patients under 18 years of age.
* Patients with severe or unstable comorbid conditions.
* Patients with active malignancy or malignancy in past 5 years (not including appropriately treated cutaneous basal and cutaneous-limited squamous cell carcinomas).
* Patients who are pregnant or breastfeeding.
* Patients with any other skin condition that prohibit or confound the ability of the investigator to interpret skin findings.
* Patients with active substance or alcohol abuse disorder; or history of substance/alcohol abuse disorder within 6 months prior to study enrollment.
* History of, or active, severe depression and/or suicidality.
* Patients with active or latent tuberculosis as determined by quant-TB baseline testing
* Patients that are taking concomitant biologics, systemics for the treatment of psoriasis and/or phototherapy.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2023-07-24 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Identify Adherence to treatment | 3 month close-out visit
  Qualitative data will be obtained from detailed, systematic interviews at 3-month follow-up to Adherence to treatment will be captured using electronic monitors that record the timing of medication dosing events and the number of pills taken at each event (based on weight of medication using Sensal Health adherence monitoring device) measured at 3 month close-out visit

SECONDARY OUTCOMES:
Psoriasis Treatment Efficacy (PASI 75) | baseline and 3 month close-out visit
  Compare psoriasis treatment outcomes between the most and least adherent patients
  The primary measure of efficacy for comparing efficacy between high vs low adherence subjects will be percent of subjects with 75% improvement in Psoriasis Area and Severity Index (PASI 75).
Psoriasis Treatment Efficacy (PASI 90) | baseline and 3 month close-out visit
  Compare psoriasis treatment outcomes between the most and least adherent patients
  The primary measure of efficacy for comparing efficacy between high vs low adherence subjects will be percent of subjects with 90% improvement in Psoriasis Area and Severity Index (PASI 90).
Psoriasis Treatment Efficacy (PASI 100) | baseline and 3 month close-out visit
  Compare psoriasis treatment outcomes between the most and least adherent patients
  The primary measure of efficacy for comparing efficacy between high vs low adherence subjects will be percent of subjects with 100% improvement in Psoriasis Area and Severity Index (PASI 100).
Disease Clarity - Investigator's Global Assessment (IGA) Scale | baseline and 3 month close-out visit
  Compare psoriasis treatment outcomes between the most and least adherent patients
  The IGA is a five-point scale is a modified tool for evaluating plaque psoriasis severity ranging from 0 to 4, where 0 indicates clear, 2 is mild, 3 is moderate, and 4 indicates severe AD. A decrease in score relates to an improvement in signs and symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Steven R Feldman, MD, PhD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest University Health Sciences Department of Dermatology, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No